CLINICAL TRIAL: NCT03774849
Title: Evaluation of the PicoWay™ Laser System With 730nm and Resolve™ Fusion Handpieces for Treatment of Benign Pigmented Lesions and Wrinkles
Brief Title: PicoWay™ 730 Resolve Fusion for Benign Pigmented Lesions and Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PWY18010
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Benign Pigmented Lesions; Facial Wrinkles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Picoway™ 532nm fractional handpiece (Experimental): Subjects will receive up to four study treatments with the PicoWay™ 532nm fractional handpiece
  Interventions: Device: PicoWay™ 730nm wavelength
- PicoWay™ 730nm wavelength (Experimental): PicoWay™ 730nm wavelength. Subjects will receive up to four study treatments with the PicoWay™ 730nm wavelength.
  Interventions: Device: PicoWay™ 532nm fractional handpiece
- PicoWay ™1064nm fractional handpiece (Experimental): Subjects will receive up to four study treatments with the PicoWay™ 1064nm fractional handpiece
  Interventions: Device: PicoWay™ 1064nm fractional handpiece

INTERVENTIONS:
Device: PicoWay™ 532nm fractional handpiece — PicoWay™ Laser System is picosecond 532/1064/785 laser
  Arms: PicoWay™ 730nm wavelength
Device: PicoWay™ 730nm wavelength — PicoWay™ Laser System is picosecond 532/1064/785 laser
  Arms: Picoway™ 532nm fractional handpiece
Device: PicoWay™ 1064nm fractional handpiece — PicoWay™ Laser System is picosecond 532/1064/785 laser
  Arms: PicoWay ™1064nm fractional handpiece

SUMMARY:
Evaluation of the PicoWay™ Laser System With 730nm and Resolve™ Fusion Handpieces for Treatment of Benign Pigmented Lesions and Wrinkles.

DETAILED DESCRIPTION:
Subjects will receive up to 4 study treatments with the PicoWay™ 730 nm laser wavelength, PicoWay™1064nm fractional handpiece and/or PicoWay™ 1064nm fractional handpiece for treatment of benign pigmented lesions or wrinkles. Subjects will return for three follow-up visit evaluations 1-month, 2-months and 3-months post final study treatment. Primary efficacy assessed by masked photographic evaluation. Optional biopsy collection for histological analysis of laser tissue effects.

ELIGIBILITY:
Inclusion Criteria

1. Willing to provide signed informed consent
2. Adults age 21 to 80
3. Fitzpatrick Skin Type (FST) I to VI
4. Presence of benign pigmented Lesions assessed at baseline as Pigment Severity Score (PSS) of "2" or higher and/or wrinkles assessed at baseline as Fitzpatrick Wrinkle Score (FWS) of "2" or higher
5. Willing to allow photographs and/or video to be taken of treated areas for the purposes of this research study
6. Willing to abstain from any other procedures for treatment of benign pigmented lesions or wrinkles in the laser treatment areas for the duration of the study including surgery, light, laser, ultrasound or radiofrequency treatments
7. Willing to abstain from use of prescription cosmetic products for treatment of benign pigmented lesions or wrinkles in the laser treatment areas for the duration of the study including injections of neurotoxins or dermal fillers, skin lightening creams, and wrinkle creams
8. Willingness to adhere to study treatment and follow-up visit schedules

Exclusion Criteria

1. Pregnant, planning pregnancy or breast feeding
2. Allergy to topical or injectable lidocaine or similar medications
3. Allergy to topical steroid or similar medications
4. Unprotected sun exposure in the six weeks prior to enrollment, or active tan in the laser treatment area
5. History of melanoma in the intended treatment area
6. History of keloid or hypertrophic scar formation
7. Use of topical or systemic retinoid therapy during the past six (6) months
8. Use of neurotoxins in the intended treatment area within the past three (3) months or throughout the duration of the study
9. Use of dermal fillers in the intended treatment area within the last six (6) months or throughout the duration of the study
10. Severe immunosuppression resulting from medications and/or a medical condition that could impair healing after treatment.
11. Open wound or infection in the intended treatment area
12. History of light induced seizure disorders
13. Dermatologic and/or cosmetic procedures in the intended treatment area(s) during the past six months
14. The subject is not suitable, in the opinion of the clinician, for participation in the study due to medical or other reasons that could compromise the study integrity or subject safety

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lowery, Study Director — Director of Clinical Affairs, Candela Corporation
Locations (1):
- Syneron Candela Institute for Excellence, Wayland, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Group A: Treatment of Benign Pigmented Lesions including dyschromia
- Group B: Group B:Wrinkles including fine lines
- Group A and B: Participants Enrolled in Both Group A and B
  Treated for Benign Pigmented lesions and Wrinkles
Period: Overall Study
Arm/Group | Group A | Group B | Group A and B
Started | 80 | 31 | 4
PicoWay 532nm | 43 | 0 | 0
PicoWay 1064nm | 1 | 31 | 0
PicoWay 730nm | 22 | 0 | 0
PicoWay 532nm and 730nm | 4 | 0 | 0
PicoWay 730nm and 1064nm | 0 | 0 | 4
Completed | 70 | 31 | 4
Not Completed | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Group A: Benign Pigmented Lesions
  Subjects will receive up to four study treatments with the PicoWay™ 532nm, 730nm, and/or 1064nm handpiece
- Group B: Group B: Wrinkles
  Subjects will receive up to four study treatments with the PicoWay™ 1064nm fractional handpiece
- Group A and B: Group A and B: BPLs and Wrinkles
  Subjects will receive up to four study treatments with the PicoWay™ 532nm, 730nm, and/or 1064nm handpiece
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group A and B | Total
Number analyzed (Participants) | 80 | 31 | 4 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9) | 56 (7) | 62 (2) | 52 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 26 | 4 | 103
  Male | 7 | 5 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 78 | 30 | 4 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 58 | 18 | 1 | 77
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 11 | 3 | 32
  More than one race | 4 | 2 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 31 | 4 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change in Wrinkles From Baseline to 12 Weeks Post-study Treatment Assessed by Blinded Photographic Evaluation Using 9-Point Fitzpatrick Wrinkle Scale
Description: 9-Point Fitzpatrick Wrinkle Scale (FWS)
  1=Fine Wrinkles to 9=Deep Wrinkles 1-3 Mild (fine textural changes with subtly accentuated skin lines) 4-6 Moderate (distinct papular elastosis [individual papules with yellow translucency under direct lighting] and dyschromia) 7-9 Severe (multipapular and confluent elastosis [thickened yellow and pallid] approaching or consistent with cutis rhomboidalis)
Time Frame: Baseline to 12-week follow-Up Visit
Population: The blinded evaluation was not conducted for the assessment of primary endpoints at this time. Investigator assessment for wrinkle reduction was conducted via internal review of 'before and after' images to assess participants treated for wrinkles but using incorrect scale, so data for this group could not be analyzed accurately. If conducted in the future, the clinical study report will be addended.
Arm/Group | Group A | Group B | Group A and B
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Subject Satisfaction Mean of Scores From 2nd Treatment Visit to Last Visit by Treatment Group Using a 5-Point Likert-type Rating Scale
Description: During the 2nd Treatment Visit and all subsequent study visits (treatment and follow-up), Subject Satisfaction Surveys were obtained from all subjects. The scale used to evaluate subject satisfaction is a Likert-type rating Scale and follows -2, -1, 0, 1, 2 for responses of Extremely Dissatisfied, Somewhat Dissatisfied, Neither Satisfied nor Dissatisfied, Somewhat Satisfied and Extremely Satisfied respectfully. The scores are stratified according to treatment group.
Time Frame: Pre-Treatment 2 at Week 6, Pre-Treatment 3 at Week 12, Pre-Treatment 4 at Week 18, 1 Month Follow-Up at Week 22, 2 Month Follow-Up at Week 26, and 3 Month Follow-Up at Week 30
Population: Some subjects received treatments on multiple areas and reported different satisfaction scores with the different areas. Thus, the units analyzed reflect the individual areas treated and not the participant. Group A&B (n=4) were double counted in this analysis because they were treated under both Group A and Group B. Group A (n=80) and Group B (n=31) is inclusive of Group A&B (n=4) subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Treated areas
Arm/Group | Group A | Group B
Number analyzed (Participants) | 80 | 31
Number analyzed (Treated areas) | 88 | 35
score on a scale
  Pre-Treatment 2 | 0.85 (0.96) | 0.65 (0.85)
  Pre-Treatment 3 | 1.16 (0.87) | 0.79 (0.84)
  Pre-Treatment 4 | 1.19 (0.88) | 0.91 (1.06)
  1 Month Follow Up | 1.13 (1.02) | 0.71 (1.24)
  2 Month Follow Up | 1.25 (1.07) | 0.72 (1.05)
  3 Month Follow Up | 1.38 (0.81) | 0.56 (1.19)

3. Primary Outcome: Change in Benign Pigmented Lesions From Baseline to 12 Weeks Post-study Treatment in Pigment Clearance Score (PCS) as Determined by Blinded Evaluators From Clinical Photography
Description: 5-Point Pigment Clearance Score (Score, Clearance %, Description)
  1. = 0-24% = Poor Response
  2. = 25-49% = Fair Response
  3. = 50-74% = Good Response
  4. = 75-94% = Excellent Response
  5. = >95% = CompleteResponse
Time Frame: Baseline to 12-week follow-Up Visit
Population: The blinded evaluation was not conducted for the assessment of primary endpoints at this time. Investigator assessment for pigment reduction was conducted via internal review of 'before and after' images to assess participants treated for benign pigmented lesions but using incorrect scale, so data for this group could not be analyzed accurately. If conducted in the future, the clinical study report will be addended.
Arm/Group | Group A | Group B | Group A and B
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline through study completion, approximately 30 weeks
Description: Candela Picoway laser system is a non-significant risk device.
Groups:
- Group A: Benign Pigmented Lesions, 532nm; Group A: Benign Pigmented Lesions, 730nm; Group A: Benign Pigmented Lesions, 1064nm; Group A: Benign Pigmented Lesions, 532nm & 730nm; Group B: Wrinkles, 1064nm: Subjects will receive up to four study treatments
- Group A and B: 730nm and 1064nm: Subjects will receive up to four study treatments. BPLs treated at 730nm, wrinkles treated at 1064nm
Arm/Group | Group A: Benign Pigmented Lesions, 532nm | Group A: Benign Pigmented Lesions, 730nm | Group A: Benign Pigmented Lesions, 1064nm | Group A: Benign Pigmented Lesions, 532nm & 730nm | Group B: Wrinkles, 1064nm | Group A and B: 730nm and 1064nm
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/22 | 0/1 | 0/4 | 0/31 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/22 | 0/1 | 0/4 | 0/31 | 0/4
Other Adverse Events (participants affected / at risk) | 13/43 | 4/22 | 0/1 | 1/4 | 2/31 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Benign Pigmented Lesions, 532nm (N=43) | Group A: Benign Pigmented Lesions, 730nm (N=22) | Group A: Benign Pigmented Lesions, 1064nm (N=1) | Group A: Benign Pigmented Lesions, 532nm & 730nm (N=4) | Group B: Wrinkles, 1064nm (N=31) | Group A and B: 730nm and 1064nm (N=4)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melasma activation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
herpetic outbreak (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
unrelated symptoms (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — headache, dizziness, aches, feeling feverish
Paradoxical Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer of nasal passage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT03774849/Prot_SAP_002.pdf